CLINICAL TRIAL: NCT02916108
Title: Interhemispheric Anterior Delta Desynchronization in Children Who Present to the Emergency Department With Acute Concussion: A Proof of Concept Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0333-16-RambamCTIL
Record Dates: First submitted 2016-09-18; First posted 2016-09-27 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Concussion, Mild Traumatic Brain Injury
Keywords: Concussion; Mild traumatic brain injury; EEG
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concussion: Study group include up to 30 children with history of concussion in the last 24 hours before admitting to emergency department.
  Reading EEG.
  Interventions: Other: Reading EEG
- Isolated limb injury: Cohort group include up to 30 children with history of isolated limb injury in the last 24 hours before admitting to emergency department.
  Reading EEG.
  Interventions: Other: Reading EEG

INTERVENTIONS:
Other: Reading EEG — EEG recording for 5 minutes (not an intervention)

SUMMARY:
Approximately 150,000 children present each year to emergency departments (EDs) in the US with concussion and many more are treated by primary care physician, or outpatient specialists.

Concussion is defined as a traumatically induced transient disturbance of brain function and involves a complex pathophysiological process. There is a variety of symptoms related to concussion, and the diagnosis of concussion requires the use of symptom-checklist. Since there is a various degree of the severity of those symptoms, the diagnosis is a subjective one and lacks sensitivity.

One major problem is that approximately one-third of the children with concussion experience ongoing somatic, cognitive, and psychological or behavioral symptoms, referred to as persistent post-concussion symptoms. A recent study that investigated the validity a 12-point PPCS risk score revealed that it had modest validity (0.71). Moreover, one of the greatest concerns is the child's schedule return to activity.

Since the basic mechanism for concussion is acceleration/ deceleration movement of axons, it is likely to be expressed in desynchronization of delta wave activity between anterior hemispheres as seen in pathological problems related to attention and/ or working memory).

The aim of this proof-of-concept study is to find-out whether interhemispheric desynchronization of delta waves (IHDD) in the anterior hemispheres can identify acute concussion in children. If the investigators find that IHDD can accurately diagnose acute concussion, a second objective will be to examine whether this index can be a useful tool in the follow up of patients with persistent post-concussion symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Study group will include children aged 11-18 years with diagnosis of acute concussion based on the RPSQ. (Eisenberg et al., 2013; Harmon et al., 2013)
* Controls will be healthy children who will be admitted to the ED due to an isolated limb injury such as laceration, contusion or fracture and are not painful. Nonverbal or non-cooperative children will be excluded from the study.

Exclusion Criteria:

* Nonverbal or non-cooperative children.
* Lack of inform consent.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A prospective case control study will be performed. The investigators will enroll patients presented to the pediatric ED of Rambam Health Care Campus (RHCC) with symptoms of acute concussion within 24 hours of mild head injury). The control group will be consisted of previously healthy children with an isolated limb injury. Study participants will be enrolled on the basis of a convenience sample.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary objective: Change in interhemispheric desynchronization of delta waves (IHDD) in the anterior hemispheres, as calculated from the sampled EEG. | One year
  Change in interhemispheric desynchronization of delta waves (IHDD) in the anterior hemispheres, as calculated from the sampled EEG.

SECONDARY OUTCOMES:
Secondary objective: Percentage of children with persistent post-concussion symptoms that display a decreased IHDD below 0.7 in the anterior hemispheres. | One year
  Percentage of children with persistent post-concussion symptoms that display a decreased IHDD below 0.7 in the anterior hemispheres.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Baron Shahaf, MD PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] DeMatteo C, McCauley D, Stazyk K, Harper J, Adamich J, Randall S, Missiuna C. Post-concussion return to play and return to school guidelines for children and youth: a scoping methodology. Disabil Rehabil. 2015;37(12):1107-12. doi: 10.3109/09638288.2014.952452. Epub 2014 Aug 21. PMID 25144831
- [Background] Eisenberg MA, Andrea J, Meehan W, Mannix R. Time interval between concussions and symptom duration. Pediatrics. 2013 Jul;132(1):8-17. doi: 10.1542/peds.2013-0432. Epub 2013 Jun 10. PMID 23753087
- [Background] Harmon KG, Drezner JA, Gammons M, Guskiewicz KM, Halstead M, Herring SA, Kutcher JS, Pana A, Putukian M, Roberts WO. American Medical Society for Sports Medicine position statement: concussion in sport. Br J Sports Med. 2013 Jan;47(1):15-26. doi: 10.1136/bjsports-2012-091941. PMID 23243113
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Baldea JD. In response to: time to re-think the Zurich Guidelines? A critique on the consensus statement on concussion in Sport&colon; the 4th International Conference on Concussion in Sport, held in Zurich, November 2012. Clin J Sport Med. 2014 Nov;24(6):521-2. doi: 10.1097/JSM.0000000000000157. No abstract available. PMID 25347264
- [Background] Potter S, Leigh E, Wade D, Fleminger S. The Rivermead Post Concussion Symptoms Questionnaire: a confirmatory factor analysis. J Neurol. 2006 Dec;253(12):1603-14. doi: 10.1007/s00415-006-0275-z. Epub 2006 Oct 24. PMID 17063314
- [Background] Shahaf G. A Possible Common Neurophysiologic Basis for MDD, Bipolar Disorder, and Schizophrenia: Lessons from Electrophysiology. Front Psychiatry. 2016 Jun 1;7:94. doi: 10.3389/fpsyt.2016.00094. eCollection 2016. PMID 27313546
- [Background] Shahaf G. Migraine as dysfunctional drive reduction: Insight from electrophysiology. Med Hypotheses. 2016 Jun;91:62-66. doi: 10.1016/j.mehy.2016.04.017. Epub 2016 Apr 11. PMID 27142146
- [Background] Shahaf G, Pratt H. Thorough specification of the neurophysiologic processes underlying behavior and of their manifestation in EEG - demonstration with the go/no-go task. Front Hum Neurosci. 2013 Jun 24;7:305. doi: 10.3389/fnhum.2013.00305. eCollection 2013. PMID 23805094
- [Background] Vargas G, Rabinowitz A, Meyer J, Arnett PA. Predictors and prevalence of postconcussion depression symptoms in collegiate athletes. J Athl Train. 2015 Mar;50(3):250-5. doi: 10.4085/1062-6050-50.3.02. Epub 2015 Feb 2. PMID 25643158
- [Background] West TA, Marion DW. Current recommendations for the diagnosis and treatment of concussion in sport: a comparison of three new guidelines. J Neurotrauma. 2014 Jan 15;31(2):159-68. doi: 10.1089/neu.2013.3031. Epub 2013 Oct 16. PMID 23879529
- [Background] Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms Among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PMID 26954410